CLINICAL TRIAL: NCT02456701
Title: Enhancing Radioiodine (RAI) Incorporation Into BRAF Mutant, RAI Refractory Thyroid Cancers With the Combination of BRAF Inhibitor Vemurafenib and Anti-ErbB3 Antibody KTN3379: A Pilot Study With a Phase 1 Run-in
Brief Title: Enhancing Radioiodine Incorporation Into BRAF Mutant Thyroid Cancers With the Combination of Vemurafenib and KTN3379
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTN3379-CL-003
Record Dates: First submitted 2015-05-20; First posted 2015-05-28 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Thyroid Cancer
Keywords: CDX3379
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination of Vemurafenib and KTN3379 (Experimental): Vemurafenib 960 mg po bid KTN3379 1000 mg IV q2weeks
  Interventions: Biological: KTN3379; Drug: vemurafenib

INTERVENTIONS:
Biological: KTN3379 — IV every 2 weeks
Drug: vemurafenib — 960 mg po bid
  Other Names: Zelboraf

SUMMARY:
This is a patient pilot study testing the hypothesis that vemurafenib with the addition of KTN3379 can restore iodine incorporation in BRAF mutant (MUT), radioiodine-refractory (RAIR) thyroid cancer patients.

DETAILED DESCRIPTION:
This is a patient pilot study testing the hypothesis that vemurafenib with the addition of KTN3379 can restore iodine incorporation in BRAF mutant (MUT), radioiodine-refractory (RAIR) thyroid cancer patients. Eligible patients with BRAF MUT, RAIR thyroid cancer will undergo human recombinant TSH (rhTSH or Thyrogen)-stimulated 124I PET/CT lesional dosimetry to quantify the baseline RAI avidity of index metastatic lesion(s). Patients will then receive vemurafenib followed by the addition of KTN3379 after which a second Thyrogen-stimulated 124I PET/CT lesional dosimetry will be performed. For patients whose tumor(s) demonstrate sufficient iodine incorporation warranting 131I therapy, Thyrogen-stimulated standard dosimetry will be performed and therapeutic 131I will be administered concurrently with vemurafenib and KTN3379. Subsequent to discontinuation of vemurafenib, tumor assessments will be conducted with serial radiologic scan(s) and thyroglobulins (scans will be performed at baseline, before 131I, 3 months (+/- 1 month) following 131I, and 6 months after 131I).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed thyroid carcinoma of follicular origin (including papillary, follicular, or poorly differentiated subtypes and their respective variants).
* Confirmation in a CLIA certified laboratory or in an FDA-approved assay that one of the patient's thyroid tumors (primary tumor, recurrent tumor, or metastasis) possesses a BRAF mutation at V600.
* Patients must have measurable disease defined by RECIST criteria 1.1.
* Tumors in previously irradiated fields may be considered measureable if there is evidence of tumor progression after radiation treatment.
* RAI-refractory disease on structural imaging
* Age ≥ 18 years.
* ECOG performance status ≤ 2
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) > 1500/mcl
  * Hemoglobin ≥ 9 g/dL
  * Platelets ≥ 100,000/mcl
  * Albumin ≥ 2.5 g/dL
  * Total bilirubin ≤ 1.5x institutional ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2x institutional ULN unless it is related to the primary disease
  * Creatinine ≤ 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) ≥ 50 mL/min OR 24-hour urine creatinine clearance ≥ 50 mL/min

Exclusion Criteria:

* Concomitant malignancies or previous malignancies treated within the past 3 years. Exception: Patients who have been disease-free for 3 years, patients with a history of completely resected non-melanoma skin cancer, and/or patients with indolent secondary malignancies, are eligible.
* Use of other investigational drugs within 28 days preceding the first dose of vemurafenib on this study.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression.
* History or evidence of cardiovascular risk including any of the following:

  * Corrected QT (QTc) interval ≥ 450 msec at baseline or history of congenital long QT syndrome or uncorrectable electrolyte abnormalities. (Patients with well controlled atrial fibrillation are exempt from this criteria.)
  * History of cerebrovascular attack or transient ischemic attack within 6 months prior to the initiation of therapy on this protocol.
  * Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10-13 (Actual); Study Completion 2016-10-13 (Actual)

PRIMARY OUTCOMES:
The number of patients with BRAF MUT, radioiodine-refractory thyroid cancer in which the combination of vemurafenib and KTN3379 can increase tumoral iodine incorporation to warrant 131I treatment | 4 to 6 weeks

SECONDARY OUTCOMES:
Safety and tolerability of the combination of vemurafenib and KTN3379 by assessing adverse events | 6 to 8 weeks

OTHER OUTCOMES:
The ORR by RECIST v1.1 criteria at 6 months following treatment with vemurafenib and KTN3379 plus 131I | 6 months
The proportion of patients alive at 6 months without disease progression by RECIST v1.1 criteria following treatment with vemurafenib and KTN3379 plus 131I | 6 months
Changes in thyroglobulin levels in patients treated with 131I | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Tchekmedyian V, Dunn L, Sherman E, Baxi SS, Grewal RK, Larson SM, Pentlow KS, Haque S, Tuttle RM, Sabra MM, Fish S, Boucai L, Walters J, Ghossein RA, Seshan VE, Knauf JA, Pfister DG, Fagin JA, Ho AL. Enhancing Radioiodine Incorporation in BRAF-Mutant, Radioiodine-Refractory Thyroid Cancers with Vemurafenib and the Anti-ErbB3 Monoclonal Antibody CDX-3379: Results of a Pilot Clinical Trial. Thyroid. 2022 Mar;32(3):273-282. doi: 10.1089/thy.2021.0565. PMID 35045748